CLINICAL TRIAL: NCT02772562
Title: A Phase II Trial of Adjuvant PROSTVAC-V/F in Subjects at High Risk for Relapse After Radical Prostatectomy
Brief Title: Adjuvant PROSTVAC-V/F in Subjects at High Risk for Relapse After Radical Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102377
Record Dates: First submitted 2016-05-03; First posted 2016-05-13 (Estimated); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROSTVAC-V/F (Experimental)
  Interventions: Biological: PROSTVAC-V/F

INTERVENTIONS:
Biological: PROSTVAC-V/F — 0.5 ml containing at least 2 x 108 Infectious Units (Inf.U) PROSTVAC-V given on day 1.
  0.5 ml containing at least 1 x 109 Inf.U PROSTVAC-F given on days 15, 28, 57, 85, 113, 141.

SUMMARY:
The purpose of this study is to see how well PROSTVAC -V/F works in stopping prostate cancer from coming back or relapsing. This study will also look at the safety of PROSTVAC-V/F.

DETAILED DESCRIPTION:
This study is for adult male patients who have recently undergone radical prostatectomy and are at high risk for relapse. The purpose of this study is to look at the effect PROSTVAC-V/F has in preventing or prolonging relapse after surgery. PROSTVAC-V/F is an investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21
2. Completed radical prostatectomy for pathologically-verified adenocarcinoma of the prostate no more than 120 days prior to start of treatment. The following procedures are acceptable: radical retropubic prostatectomy (RRP), laparoscopic radical prostatectomy (with or without robotic assistance; LAPD), radical perineal prostatectomy (RPP).
3. Post-operative PSA <0.2ng/mL by 120 days after prostatectomy
4. Must have one or more of the following:

   * pT3b or pT4 primary tumor
   * Gleason score 8-10
   * pN1 lymph node disease
   * positive surgical margins
   * pre-operative PSA of > 10ng/mL
   * presence of any tertiary Gleason 5 component on the prostatectomy pathology report.

   Note: Patients with pT3a disease who lack one of the above criteria, and who refuse adjuvant radiation, may also be enrolled.
5. ECOG performance status 0-1
6. Adequate hematologic, renal, liver function per parameters in Table 1
7. Subject of fathering potential must agree to use an adequate method of contraception to avoid conception throughout the study and for at least 4 weeks after the last dose of study drug to minimize the risk of pregnancy.
8. Subjects must have had a negative bone scan, and CT of abdomen and pelvis within 16 weeks prior to registration. Additional forms of imaging (Prostascint scan, MRI) may be substituted for a CT scan of the abdomen and pelvis if clinically indicated.

Exclusion Criteria:

1. Pure small cell carcinoma of the prostate
2. Radiographically-demonstrable metastases at any time prior to the time of enrollment
3. Diagnosis of cancer requiring systemic therapy in the past 5 years
4. Presence of any major medical condition which, in the opinion of the investigator, precludes participation in the study
5. Neoadjuvant or adjuvant therapy of any kind
6. Chronic administration (defined as daily or every other day for continued use > 14 days) of systemic glucocorticoids within 28 days of the first planned dose of PROSTVAC-V/F. Use of inhaled steroids, nasal sprays, and all topical preparations (creams, solutions, gels, ointments, etc.) for up to 5% of the body surface area is allowed.
7. Use of systemic immunosuppressant agents including anti-metabolites, glucocorticoids, TNF antagonists, antibodies to IL6 or IL6R, calcineurin inhibitors, mTOR antagonists
8. Prior history of serious toxicity or a systemic reaction to vaccinia immunization such as myopericarditis progressive vaccinia infection, or eczema vaccinatum.
9. Inflammatory or exfoliative skin diseases such as eczema, psoriasis that disrupt epidermis
10. Active infections requiring systemic therapy
11. Serologic evidence of HIV/AIDS.
12. Positive hepatitis C serology or active hepatitis B infection.
13. History of allergy to eggs, egg products, aminoglycoside antibiotics
14. History of myocardial disease, such as myocarditis, cardiomyopathy, congestive heart failure, ischemic cardiomyopathy
15. Prior solid organ or stem cell transplant
16. History of or active autoimmune disease (e.g., autoimmune neutropenia, thrombocytopenia, or hemolytic anemia, systemic lupus, localized lupus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, or Addison's disease). Persons with vitiligo, Hashimoto's thyroiditis, or Graves disease are not excluded.
17. Vaccination with live attenuated vaccine within 28 days prior to day 1 of PROSTVAC-V/F administration or vaccination with a killed vaccine within 14 days prior to day 1 of PROSTVAC-V/F.
18. Inability to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination or until the vaccination site heals completely: (a) children ≤ 3 years of age; (b) pregnant or nursing women; (c) individuals with prior or concurrent extensive eczema or other eczemoid skin disorders; or (d) immunocompromised individuals, such as those with HIV.
19. Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including Follow-Up), or would interfere with the evaluation of the trial endpoints.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PROSTVAC-V/F
Started | 33
Completed | 31
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | PROSTVAC-V/F
Number analyzed (Participants) | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.0 [61 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Relapse-Free Survival (RFS) at 2 Years Post-Prostatectomy
Description: RFS is defined as the absence of relapse (PSA ≥ 0.2 ng/mL confirmed >30 days later, radiographic metastasis, initiation of new prostate cancer therapy, or death) at 2 years after prostatectomy. The measure represents the proportion of participants who remain relapse-free at 24 months post-surgery.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | PROSTVAC-V/F
Number analyzed (Participants) | 31
Proportion of participants | 0.352 (.97) [0.154 to 0.55]

2. Secondary Outcome: Comparison of Observed vs. Predicted RFS
Description: A secondary endpoint will be a comparison of the observed RFSs with the predicted ("virtual") RFS for the same patients based on clinical and pathologic information collected at baseline. The observed RFSs of the treated subjects are compared with the predicted RFSs as if the same subjects had not been treated. The comparison is performed using the logrank test of the observed and predicted RFSs. These represent the estimated RFSs for patients with those clinical characteristics if they did not receive any adjuvant therapy.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | PROSTVAC-V/F
Number analyzed (Participants) | 31
proportion of participants | .352 [.154 to .55]

3. Secondary Outcome: Observed Relapse Free Survival (RFS) With the RFSs of a Historical Comparison Group of MUSC Prostatectomy Patients.
Description: No participants were analyzed for this outcome. Although the outcome was pre-specified in the protocol, the study was terminated early and the planned analysis comparing observed relapse-free survival (RFS) to a historical control group could not be completed. Additionally, the analysis population for this outcome was not clearly defined at the time of study closure, and no summary data were generated.
Time Frame: 2 years
Population: No participants were analyzed for this outcome. Although the outcome was pre-specified in the protocol, the study was terminated early and the planned analysis comparing observed relapse-free survival (RFS) to a historical control group could not be completed. Additionally, the analysis population for this outcome was not clearly defined at the time of study closure, and no summary data were generated.
Measure: Count of Participants; unit: Participants
Arm/Group | PROSTVAC-V/F
Number analyzed (Participants) | 0
Participants | 0

4. Secondary Outcome: Associations Between RFS Values and Research Specimen
Description: While most participants were assessed at the scheduled time points, no usable samples due to issues such as hemolysis, insufficient volume, or improper storage conditions rendered them unusable for the planned immunologic assays. No data are available for this outcome measure due to these technical limitations.
Time Frame: 2 years
Population: While most participants were assessed at the scheduled time points, no usable samples due to issues such as hemolysis, insufficient volume, or improper storage conditions rendered them unusable for the planned immunologic assays. No data are available for this outcome measure due to these technical limitations.
Measure: Count of Participants; unit: Participants
Arm/Group | PROSTVAC-V/F
Number analyzed (Participants) | 0
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | PROSTVAC-V/F
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROSTVAC-V/F (N=32)
Myocardial Infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROSTVAC-V/F (N=32)
Injection site reaction (General) | 13
Fatigue (General) | 6
Flu like symptoms (General) | 6
Fever (General) | 4
Injection site pain (General) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Other Vomiting (Gastrointestinal disorders) | 3
Increased Alt (Blood) | 2
Increased Ast (Blood) | 2
Chills (General) | 2
Edema limbs (General) | 2
Other Malaise (General) | 2
Other Depression (Psychiatric disorders) | 2
Other Urinary Frequency (Renal and urinary disorders) | 2
Other Pruritus (Skin) | 2
Other Alkaline Phosphotase Increased (Blood) | 1
Other Hemoglobinopathy (Blood) | 1
Other Hypertension (Cardiac disorders) | 1
Other Pounding Sensation; Right Ear (Ear) | 1
Other Constipation (Gastrointestinal disorders) | 1
Other Dyspepsia (Gastrointestinal disorders) | 1
Other Gastric Hemorrhage (Gastrointestinal disorders) | 1
Other Hypokalemia (General) | 1
Other Anemia (Immune) | 1
Other Sinusitis (Infections and infestations) | 1
Other Stye (Infections and infestations) | 1
Other Uri (Infections and infestations) | 1
Other Rib Fracture (Injury) | 1
Other Weight Loss (Investigations) | 1
Other Hypocarbia (Metabolism) | 1
Other Hypophosphatemia (Metabolism) | 1
Other Aches (Musculoskeletal and connective tissue disorders) | 1
Other Back Pain (Musculoskeletal and connective tissue disorders) | 1
Other Breast Soreness (Musculoskeletal and connective tissue disorders) | 1
Other Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Other Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 1
Other Joint Pain (Musculoskeletal and connective tissue disorders) | 1
Other Leg Cramping In Left Leg (Musculoskeletal and connective tissue disorders) | 1
Other Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Other Stiffness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Other Agitation (Psychiatric disorders) | 1
Other Bladder Spasms (Renal and urinary disorders) | 1
Other Dysuria (Renal and urinary disorders) | 1
Other Testicular Pain (Left) (Reproductive) | 1
Other Cough (Respiratory, thoracic and mediastinal disorders) | 1
Other Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Other Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Other Left Chest Dermatomal Erythematous Papules And Erosions (Skin) | 1
Other Lesion L Middle Finger (Skin) | 1
Other Lesion L Knee (Skin) | 1
Other Lesion Lower Lip (Skin) | 1
Other New Bump On Left Arm (Skin) | 1
Other Rash (Skin) | 1
Other Dental Caries (Abscessed Tooth Extraction) (Surgical and medical procedures) | 1
Other Incisional Hernia (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT02772562/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT02772562/ICF_001.pdf